CLINICAL TRIAL: NCT05028218
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of TQB3824 in Subjects With Advanced Cancer
Brief Title: A Clinical Study of TQB3824 in Subjects With Advanced Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3824-I-01
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3824 tablets (Experimental): TQB3824 tablets orally administrated orally on Days 1-21 of each 21-day treatment cycle. Dose escalation of TQB3824 will be based on evaluation of clinical safety and tolerability and guided by accumulating PK data
  Interventions: Drug: TQB3824 tablets

INTERVENTIONS:
Drug: TQB3824 tablets — TQB3824 is a CDC7 inhibitor, which plays important roles in the maintenance of DNA replication forks and DNA damage response pathways.

SUMMARY:
TQB3824 blocks function of a specific protein called Cell Division Cycle 7 (CDC7) kinase in the human body, which plays important roles in the maintenance of DNA replication forks and DNA damage response pathways. This study will evaluate the safety, tolerability and pharmacokinetics of TQB3824.

ELIGIBILITY:
Inclusion Criteria:

1. Understood and signed an informed consent form;
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
3. Life expectancy >=3 months;
4. Progressed after standard treatment or no standard treatment with an established survival benefit is available;
5. Adequate organ/system function;
6. Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after study is stopped; male patients should agree to use contraception during the study period and for at least 6 months after study is stopped.

Exclusion Criteria:

1. Diagnosed and/or treated additional malignancy within 3 years before the first dose;
2. With factors affecting oral medication;
3. Toxicity that is >=Grade 2 caused by previous cancer therapy;
4. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before the first dose;
5. Arterial thromboembolism and/or venous thromboembolism within 6 months;
6. A history of psychotropic drug abuse or have a mental disorder;
7. Any severe and/or uncontrolled disease;
8. Has received surgery, chemotherapy, radiotherapy or other anticancer therapies 4 weeks before the first dose;
9. Has received Chinese patent medicines with anti-tumor indications that National Medical Products Administration (NMPA) approved within 2 weeks before the first dose;
10. Has received CDC7 inhibitors;
11. Pleural effusion, pericardial effusion or ascites that cannot be controlled and need repeated drainage;
12. Brain metastases ;
13. Has participated in other clinical studies within 4 weeks before the first dose;
14. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | up to 18 months
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Maximum Tolerated Dose (MTD) | up to 18 months
  The maximum Dose at which less than 33% subjects experiencing DLT
Recommended Phase II Dose (RP2D) | up to 18 months
  RP2D will be based on evaluation of clinical safety and tolerability and guided by accumulating PK data

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | up to 18 months
  Concentration Uncer Curve
Maximum (peak) plasma drug concentration (Cmax) | up to 18 months
  Maximum plasma concentration of drug
Time to reach maximum(peak )plasma concentration following drug administration (Tmax) | up to 18 months
  Time to Reach the Maximum Plasma Concentration
Overall response rate (ORR) | Baseline up to 12 months
  The sum of percentage of participants with complete response rate and partial response rate
Disease Control Rate (DCR ) | Baseline up to 12 months
  percentage of participants with complete response (CR), partial response (PR) plus stable disease (SD)
Duration of Response (DOR) | Baseline up to 12 months
  the time from the date of first documentation of a CR or PR to the date of first documentation of tumor progression
Progression-free survival (PFS) | Baseline up to 12 months
  Time from the first dose to the first documentation of PD or death from any cause, whichever occurs first
Overall survival (OS) | Baseline up to 12 months
  the time from start of study treatment to date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institution & Hospital, Tianjin, Tianjin Municipality, China